CLINICAL TRIAL: NCT01999114
Title: A Randomized, Triple-blind, Placebo- and Positive-Controlled, Parallel Group Study of the Effect of Buprenorphine Delivered by the Buprenorphine Transdermal System (BTDS) at Doses up to 80 mcg/Hour and Naltrexone on ECG Intervals in Healthy Adult Subjects
Brief Title: The Effect of Buprenorphine Delivered by Buprenorphine Transdermal System (BTDS) at Doses up to 80 Micrograms/Hour (mcg/hr) and Naltrexone on Electrocardiogram (ECG) Intervals in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BUP1025
Record Dates: First submitted 2013-11-19; First posted 2013-12-03 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-02

CONDITIONS: ECG Effects
Keywords: Healthy subjects; Opioid; Transdermal; ECG
MeSH Terms: interventions — Buprenorphine; Naltrexone; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- BTDS (Experimental): Buprenorphine transdermal patches 10, 40 (2 x 20), and 80 (4 x 20) mcg/hr
  Interventions: Drug: Buprenorphine transdermal patch
- BTDS with naltrexone (Experimental): Buprenorphine transdermal patches 10, 40 (2 x 20), and 80 (4 x 20) mcg/hr and naltrexone 50 mg tablets
  Interventions: Drug: Buprenorphine transdermal patch; Drug: Naltrexone tablet
- Naltrexone (Active Comparator): Naltrexone 50 mg tablets
  Interventions: Drug: Naltrexone tablet
- Placebo (Placebo Comparator): Matching placebo for transdermal patches and/or naltrexone tablets and/or moxifloxacin tablets
  Interventions: Drug: Placebos (for TDS and for naltrexone and for moxifloxacin)
- Moxifloxacin (Active Comparator): Moxifloxacin 400-mg tablets
  Interventions: Drug: Moxifloxacin tablet

INTERVENTIONS:
Drug: Buprenorphine transdermal patch — Buprenorphine patch applied transdermally
  Other Names: Butrans
  Arms: BTDS; BTDS with naltrexone
Drug: Naltrexone tablet — Naltrexone tablet; 1 tablet taken orally every 12 hours
  Other Names: ReVia
  Arms: BTDS with naltrexone; Naltrexone
Drug: Placebos (for TDS and for naltrexone and for moxifloxacin) — Matching placebos
  Arms: Placebo
Drug: Moxifloxacin tablet — Moxifloxacin tablet; 1 tablet taken orally on Days 6, 13 and 17
  Other Names: Avelox®
  Arms: Moxifloxacin

SUMMARY:
The purpose of this study is to evaluate the ECG effects of 10, 40, and 80 mcg/hr buprenorphine delivered by BTDS alone, or by BTDS dosed with naltrexone, relative to placebo in healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Males and females aged 18 to 55, inclusive.
* Body weight ranging from 50 to 100 kilograms (kg) (110 to 220 lbs) and body mass index (BMI) ranging from 18 to 30 (kg/m2), inclusive.
* Healthy and free of significant abnormal findings as determined by medical history, physical examination, clinical laboratory values, vital signs, and resting 12-lead ECG.
* Females of child-bearing potential must be using an adequate and reliable method of contraception (ie, barrier with additional spermicidal foam or jelly, intra-uterine device, hormonal contraception). Females who are postmenopausal must have been postmenopausal ≥ 1 year and have elevated serum follicle stimulating hormone (FSH).
* Willing to eat the food supplied during the study.
* Willing to refrain from strenuous exercise during the entire study. Subjects will not begin a new exercise program nor participate in any unusually strenuous physical exertion.
* All 8 anatomical transdermal system (TDS) application sites (upper back, upper chest, upper outer arm, or lateral thorax) must be acceptable for study use.

Exclusion Criteria:

* Females who are pregnant (positive beta human chorionic gonadotropin test) or lactating.
* Current or recent (within 5 years) history of drug or alcohol abuse.
* History or any current conditions that might interfere with drug absorption (transdermal or gastrointestinal), distribution, metabolism or excretion.
* Use of an opioid-containing medication in the past 30 days preceding the initial dose in this study.
* Known allergy to buprenorphine, any excipient of BTDS, opioids, psychotropic or hypnotic drugs, and/or moxifloxacin or any member of the quinolone class drugs.
* Any history of frequent nausea or emesis regardless of etiology.
* Any history of seizures or head trauma with sequelae.
* Participation in a clinical drug study during the 30 days preceding the initial dose in this study.
* Any significant illness during the 30 days preceding the initial dose in this study.
* Use of any medication including thyroid hormonal therapy (hormonal contraception and hormonal replacement therapy in the form of estrogen with or without progestin is allowed), vitamins, herbal and/or mineral supplements during the 7 days preceding the initial dose.
* Any personal or family history of prolonged QT interval or disorders of cardiac rhythm.
* Abnormal cardiac conditions including hypertension.
* Abnormal cardiac condition denoted by any of the following:

  * QTcF interval > 450 milliseconds (msec)
  * PR interval > 240 msec or QRS > 110 msec
  * Evidence of second- or third-degree atrioventricular (AV) block
  * Pathological Q-waves (defined as Q-wave >40 msec or depth > 0.5 mV)
  * Evidence of ventricular pre-excitation, complete left bundle branch block, right bundle branch block (RBBB), or incomplete RBBB
  * With a resting heart rate outside the range of 45 to 85 beats per minute (bpm)
* Abnormalities on physical examination, vital signs, ECG, or clinical laboratory values, unless those abnormalities were judged clinically insignificant by the investigator.
* Oxygen saturation (SpO2) ≤ 94% as measured by pulse oximetry.
* Refusal to abstain from caffeine or xanthine containing beverages entirely during confinement.
* Refusal to abstain from consumption of alcoholic beverages 48 hours prior to initial study drug administration and any time during study.
* History of smoking or use of nicotine products within 45 days of study drug administration or a positive urine cotinine test
* Blood or blood products donated within 30 days prior to study drug administration or anytime during the study.
* Positive results of urine drug screen or alcohol screen.
* Positive results of hepatitis B surface antigen (HBsAg), hepatitis C antibody (anti-HCV).
* Positive naloxone challenge test.
* Presence of Gilbert's Syndrome, or any known hepatobiliary abnormalities.
* The investigator believes the subject to be unsuitable for reason(s) not specifically stated in the exclusion criteria.
* Subjects who have allergies or other contraindications to transdermal systems or patch adhesives.
* Clinically significant history of allergic reaction to wound dressings or elastoplast.
* Subjects with a dermatological disorder at any relevant patch application site that precludes proper placement and/or rotation of patch.
* Taking antihistamines within 72 hours prior to dosing or systemic or topical corticosteroids within 3 weeks prior to dosing.
* Subjects will not allow hair to be removed at the proposed patch application site which may prevent proper placement of the patch.
* Subjects for whom a proper assessment of possible application site reactions would be confounded by local skin conditions.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 328 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States

REFERENCES:
- [Result] Harris SC, Morganroth J, Ripa SR, Thorn MD, Colucci S. Effects of buprenorphine on QT intervals in healthy subjects: results of 2 randomized positive- and placebo-controlled trials. Postgrad Med. 2017 Jan;129(1):69-80. doi: 10.1080/00325481.2017.1270156. PMID 27927048

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject First Visit: 15-March-2012; Last Subject Last Visit: 10-October-2012. The study was conducted at 1 medical/research site in the United States.
Pre-assignment Details: Healthy adult subjects
Groups:
- BTDS: Buprenorphine transdermal patches 10, 40 (2 x 20) and 80 (4 x 20) mcg/hr
  Buprenorphine transdermal patch: Buprenorphine patch applied transdermally
- BTDS With Naltrexone: Buprenorphine transdermal patches 10, 40 (2 x 20) and 80 (4 x 20) mcg/hr and naltrexone 50 mg tablets
  Buprenorphine transdermal patch: Buprenorphine patch applied transdermally
  Naltrexone tablet: Naltrexone tablet; 1 tablet taken orally every 12 hours
- Placebo: Matching placebo for transdermal patches and/or naltrexone tablets and/or moxifloxacin tablets
  Placebos (for BTDS and for naltrexone and for moxifloxacin): Matching placebos
Period: Overall Study
Arm/Group | BTDS | BTDS With Naltrexone | Naltrexone | Moxifloxacin | Placebo
Started | 66 | 66 | 66 | 65 | 65
Completed | 58 | 59 | 61 | 62 | 61
Not Completed | 8 | 7 | 5 | 3 | 4
Not completed — Adverse Event | 8 | 7 | 2 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Administrative | 0 | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BTDS | BTDS With Naltrexone | Naltrexone | Moxifloxacin | Placebo | Total
Number analyzed (Participants) | 66 | 66 | 66 | 65 | 65 | 328
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (9.27) | 31.6 (8.97) | 34.0 (10.14) | 35.0 (10.03) | 33.0 (10.48) | 33.4 (9.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 22 | 29 | 23 | 127
  Male | 40 | 39 | 44 | 36 | 42 | 201
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 0 | 2
  Asian | 1 | 3 | 0 | 1 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 22 | 21 | 22 | 26 | 24 | 115
  White | 41 | 41 | 44 | 38 | 40 | 204
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Time-matched Change From Baseline in QT Data Corrected for Heart Rate (QTc), Placebo-corrected, Based on an Individual Correction (QTcI) Method (ΔΔQTcI)
Description: The effects of 10 mcg/hr buprenorphine (Day 6) delivered by BTDS alone, or by BTDS dosed with naltrexone, and naltrexone alone on cardiac repolarization, were assessed based on the corrected QT interval since HR inversely affects QT duration. The time-matched analysis was conducted as the primary endpoint as recommended by ICH E14, with the 2-sided 90% confidence interval for each treatment at each time point showing the placebo- and baseline-corrected (ΔΔ) analysis for QTcI. The effect of BTDS 10 on QT intervals was compared with the moxifloxacin-positive control after placebo and baseline correction.
Time Frame: Baseline to Day 6
Population: The full analysis for ECG population was the group of subjects who were randomized, received at least 1 dose of study drug, and had at least 1 time-matched baseline and 1 on-treatment ECG.
  The placebo treatment group is not presented; however, the placebo data were used as a correction factor for these time-matched analyses.
Measure: Mean (90% Confidence Interval); unit: milliseconds (msec)
Groups:
- BTDS Only (Placebo-corrected ΔΔQTcI): BTDS 10 mcg/hr
- BTDS With Naltrexone (Placebo-corrected ΔΔQTcI): BTDS 10 mcg/hr and naltrexone 50 mg tablets
- Naltrexone Alone (Placebo-corrected ΔΔQTcI): Naltrexone 50 mg tablets
- Moxifloxacin (Placebo-corrected ΔΔQTcI): Moxifloxacin 400 mg tablet (positive control)
Arm/Group | BTDS Only (Placebo-corrected ΔΔQTcI) | BTDS With Naltrexone (Placebo-corrected ΔΔQTcI) | Naltrexone Alone (Placebo-corrected ΔΔQTcI) | Moxifloxacin (Placebo-corrected ΔΔQTcI)
Number analyzed (Participants) | 66 | 63 | 65 | 64
milliseconds (msec) | 3.36 [1.09 to 5.63] | 5.37 [2.70 to 8.03] | 4.34 [2.21 to 6.48] | 11.90 [8.82 to 14.97]

2. Primary Outcome: The Maximum Time-matched Change From Baseline in QT Data Corrected for Heart Rate (QTc), Placebo-corrected, Based on an Individual Correction (QTcI) Method (ΔΔQTcI)
Description: The effects of 40 mcg/hr buprenorphine (Day 13) delivered by BTDS alone, or by BTDS dosed with naltrexone, and naltrexone alone on cardiac repolarization, were assessed based on the corrected QT interval since HR inversely affects QT duration. The time-matched analysis was conducted as the primary endpoint as recommended by ICH E14, with the 2-sided 90% confidence interval for each treatment at each time point showing the placebo- and baseline-corrected (ΔΔ) analysis for QTcI. The effect of BTDS 40 on QT intervals was compared with the moxifloxacin-positive control after placebo and baseline correction.
Time Frame: Baseline to Day 13
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: msec
Groups:
- BTDS Only (Placebo-corrected ΔΔQTcI): BTDS 40 mcg/hr
- BTDS With Naltrexone (Placebo-corrected ΔΔQTcI): BTDS 40 mcg/hr and naltrexone 50 mg tablets
- Moxifloxacin (Placebo-corrected ΔΔQTcI): Moxifoxacin 400 mg tablet (positive control)
Arm/Group | BTDS Only (Placebo-corrected ΔΔQTcI) | BTDS With Naltrexone (Placebo-corrected ΔΔQTcI) | Naltrexone Alone (Placebo-corrected ΔΔQTcI) | Moxifloxacin (Placebo-corrected ΔΔQTcI)
Number analyzed (Participants) | 63 | 63 | 64 | 64
msec | 9.16 [6.52 to 11.81] | 5.12 [2.26 to 7.97] | 1.81 [-0.70 to 4.33] | 10.68 [7.06 to 14.30]

3. Primary Outcome: The Maximum Time-matched Change From Baseline in QT Data Corrected for Heart Rate (QTc), Placebo-corrected, Based on an Individual Correction (QTcI) Method (ΔΔQTcI)
Description: The effects of 80 mcg/hr buprenorphine (Day 17) delivered by BTDS alone, or by BTDS dosed with naltrexone, and naltrexone alone on cardiac repolarization, were assessed based on the corrected QT interval since HR inversely affects QT duration. The time-matched analysis was conducted as the primary endpoint as recommended by ICH E14, with the 2-sided 90% confidence interval for each treatment at each time point showing the placebo- and baseline-corrected (ΔΔ) analysis for QTcI. The effect of BTDS 80 on QT intervals was compared with the moxifloxacin-positive control after placebo and baseline correction.
Time Frame: Baseline to Day 17
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: msec
Groups:
- BTDS Only (Placebo-corrected ΔΔQTcI): BTDS 80 mcg/hr
- BTDS With Naltrexone (Placebo-corrected ΔΔQTcI): BTDS 80 mcg/hr and naltrexone 50 mg tablets
Arm/Group | BTDS Only (Placebo-corrected ΔΔQTcI) | BTDS With Naltrexone (Placebo-corrected ΔΔQTcI) | Naltrexone Alone (Placebo-corrected ΔΔQTcI) | Moxifloxacin (Placebo-corrected ΔΔQTcI)
Number analyzed (Participants) | 58 | 62 | 63 | 64
msec | 11.46 [8.78 to 14.14] | 4.47 [1.71 to 7.23] | 1.50 [-1.15 to 4.15] | 10.78 [7.20 to 14.35]

4. Secondary Outcome: QTcF and QTcB for Historical Purposes, PR Interval, QRS Interval, and Uncorrected QT Interval
Description: Mean change from baseline for the BTDS 10 mcg/hr dose on Day 6, presented as time-averaged mean change from baseline for BTDS only, BTDS with naltrexone, naltrexone alone, moxifloxacin, and placebo.
Time Frame: Baseline to Day 6
Population: The full analysis for ECG population was the group of subjects who were randomized, received at least 1 dose of study drug, and had at least 1 time-matched baseline and 1 on-treatment ECG.
Measure: Mean (Standard Deviation); unit: msec
Groups:
- BTDS Only: BTDS 10 mcg/hr
- BTDS With Naltrexone: BTDS 10 mcg/hr and naltrexone 50 mg tablets
- Naltrexone Alone: Naltrexone 50 mg tablets
- Moxifloxacin: Moxifloxacin 400 mg tablet (positive control)
Arm/Group | BTDS Only | BTDS With Naltrexone | Naltrexone Alone | Moxifloxacin | Placebo
Number analyzed (Participants) | 66 | 63 | 65 | 64 | 64
msec
  QTcF | -0.1 (5.9) | 2.9 (8.7) | 1.5 (4.6) | 6.9 (5.1) | -0.8 (5.4)
  QTcB | -0.3 (6.1) | 1.5 (6.6) | 0.9 (5.4) | 9.1 (5.2) | 0.5 (7.0)
  PR | 4.7 (7.2) | 2.4 (5.0) | 2.1 (4.2) | 0.3 (6.1) | 0.6 (4.4)
  QRS | 0.4 (2.1) | 0.7 (1.9) | 0.6 (1.4) | -0.2 (1.9) | 0.0 (1.5)
  QT | 0.3 (11.2) | 5.6 (22.1) | 2.6 (8.8) | 2.6 (11.9) | -3.4 (8.6)

5. Secondary Outcome: Heart Rate (HR)
Description: as for outcome 4
Time Frame: Baseline to Day 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | BTDS Only | BTDS With Naltrexone | Naltrexone Alone | Moxifloxacin | Placebo
Number analyzed (Participants) | 66 | 63 | 65 | 64 | 64
bpm | -0.1 (3.8) | -1.3 (6.8) | -0.5 (2.9) | 2.0 (4.1) | 1.3 (3.3)

6. Secondary Outcome: QTcF and QTcB for Historical Purposes, PR Interval, QRS Interval, and Uncorrected QT Interval
Description: Mean change from baseline for the BTDS 40 mcg/hr dose on Day 13, presented as time-averaged mean change from baseline for BTDS only, BTDS with naltrexone, naltrexone alone, moxifloxacin, and placebo.
Time Frame: Baseline to Day 13
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: msec
Groups:
- BTDS Only: BTDS 40 mcg/hr
- BTDS With Naltrexone: BTDS 40 mcg/hr and naltrexone 50 mg tablets
- Moxifloxacin: Moxifloxacin 400 mg tablets
Arm/Group | BTDS Only | BTDS With Naltrexone | Naltrexone Alone | Moxifloxacin | Placebo
Number analyzed (Participants) | 63 | 63 | 64 | 64 | 62
msec
  QTcF | 5.0 (7.8) | 1.1 (9.6) | -1.3 (6.2) | 5.6 (6.6) | -1.6 (6.2)
  QTcB | 6.3 (8.8) | -1.1 (8.0) | -2.2 (6.8) | 8.0 (7.0) | 0.2 (7.2)
  PR | 4.5 (8.7) | 4.4 (5.9) | 3.2 (9.1) | 1.3 (6.6) | 2.0 (5.5)
  QRS | 0.2 (2.8) | 0.9 (2.4) | 1.3 (2.0) | -0.2 (2.6) | 0.3 (1.8)
  QT | 2.4 (16.0) | 5.5 (20.8) | 0.4 (11.3) | 0.9 (13.8) | -5.1 (12.6)

7. Secondary Outcome: Heart Rate (HR)
Description: as for outcome 6
Time Frame: Baseline to Day 13
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | BTDS Only | BTDS With Naltrexone | Naltrexone Alone | Moxifloxacin | Placebo
Number analyzed (Participants) | 63 | 63 | 64 | 64 | 62
bpm | 1.3 (5.9) | -1.9 (6.3) | -0.8 (3.7) | 2.3 (5.0) | 1.6 (4.5)

8. Secondary Outcome: QTcF and QTcB for Historical Purposes, PR Interval, QRS Interval, and Uncorrected QT Interval
Description: Mean change from baseline for the BTDS 80 mcg/hr dose on Day 17, presented as time-averaged mean change from baseline for BTDS only, BTDS with naltrexone, naltrexone alone, moxifloxacin, and placebo.
Time Frame: Baseline to Day 17
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: msec
Groups:
- BTDS Only: BTDS 80 mcg/hr
- BTDS With Naltrexone: BTDS 80 mcg/hr and naltrexone 50 mg tablets
Arm/Group | BTDS Only | BTDS With Naltrexone | Naltrexone Alone | Moxifloxacin | Placebo
Number analyzed (Participants) | 58 | 62 | 63 | 64 | 62
msec
  QTcF | 9.0 (7.6) | 1.8 (8.6) | -0.8 (7.4) | 6.7 (6.4) | -0.4 (6.6)
  QTcB | 10.4 (9.0) | -0.8 (8.7) | -1.7 (7.9) | 9.3 (7.7) | 1.2 (7.6)
  PR | 5.4 (8.9) | 5.8 (5.5) | 4.3 (5.7) | 3.8 (10.9) | 3.0 (5.3)
  QRS | 0.4 (3.0) | 1.5 (2.3) | 1.3 (1.9) | 0.2 (2.8) | 0.6 (1.6)
  QT | 6.1 (13.9) | 7.1 (17.1) | 0.8 (12.6) | 1.4 (11.9) | -3.7 (11.7)

9. Secondary Outcome: Heart Rate (HR)
Description: as for outcome 8
Time Frame: Baseline to Day 17
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | BTDS Only | BTDS With Naltrexone | Naltrexone Alone | Moxifloxacin | Placebo
Number analyzed (Participants) | 58 | 62 | 63 | 64 | 62
bpm | 1.3 (4.9) | -2.4 (5.6) | -0.8 (3.9) | 2.5 (4.4) | 1.5 (4.0)

10. Secondary Outcome: ECG Morphology
Description: Morphological analyses were performed with regard to the digital ECG waveform interpretation as defined by a central ECG laboratory's cardiologist blinded to the study treatment. Changes from baseline to each day of treatment were evaluated separately. Any T-U wave complex that suggested an abnormal form compatible with an effect on cardiac repolarization was noted. New ECG morphological onset changes were presented as the percentage of subjects meeting the "new" criterion ("new" meant not present on any baseline ECG and became present on at least 1 on-treatment ECG) for the following variables:
  * Second degree heart block
  * Third degree heart block
  * Complete right bundle branch block (RBBB)
  * Complete left bundle branch block (LBBB)
  * ST segment changes (elevation and depression separately)
  * T-wave abnormalities (negative T waves only)
  * Myocardial infarction (MI) pattern
  * Any new abnormal U waves
Time Frame: Baseline to Day 6
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | BTDS Only | BTDS With Naltrexone | Naltrexone Alone | Moxifloxacin | Placebo
Number analyzed (Participants) | 66 | 63 | 65 | 64 | 64
Participants
  New abnormal U waves | 0 | 0 | 0 | 0 | 0
  New T wave (negative) inverted | 1 | 0 | 1 | 0 | 0
  New ST segment depression changes | 0 | 0 | 0 | 1 | 0
  New ST segment elevation changes | 0 | 0 | 0 | 0 | 0
  New complete RBBB & LBBB | 0 | 0 | 0 | 0 | 0
  New MI | 0 | 0 | 0 | 0 | 0
  New 2nd or 3rd degree heart block | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: ECG Morphology
Description: as for outcome 10
Time Frame: Baseline to Day 13
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | BTDS Only | BTDS With Naltrexone | Naltrexone Alone | Moxifloxacin | Placebo
Number analyzed (Participants) | 63 | 63 | 64 | 64 | 62
Participants
  New abnormal U waves | 1 | 0 | 0 | 0 | 0
  New T wave (negative) inverted | 0 | 1 | 1 | 1 | 0
  New ST segment depression changes | 0 | 1 | 0 | 1 | 0
  New ST segment elevation changes | 0 | 0 | 0 | 0 | 1
  New complete RBBB & LBBB | 0 | 0 | 0 | 0 | 0
  New MI | 0 | 0 | 0 | 0 | 0
  New 2nd or 3rd degree heart block | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: ECG Morphology
Description: as for outcome 10
Time Frame: Baseline to Day 17
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | BTDS Only | BTDS With Naltrexone | Naltrexone Alone | Moxifloxacin | Placebo
Number analyzed (Participants) | 58 | 62 | 63 | 64 | 62
Participants
  New abnormal U waves | 0 | 0 | 0 | 0 | 0
  New T wave (negative) inverted | 0 | 1 | 0 | 1 | 0
  New ST segment depression changes | 1 | 0 | 0 | 1 | 0
  New ST segment elevation changes | 0 | 0 | 0 | 0 | 0
  New complete RBBB & LBBB | 0 | 0 | 0 | 0 | 0
  New MI | 0 | 0 | 0 | 0 | 0
  New 2nd or 3rd degree heart block | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were reported from start of study participation through the period beyond study completion; AEs were reported through 7 days and SAEs through 30 days after last study drug dose, or until last study visit, whichever was later.
Description: AEs were learned of through spontaneous reports or subject interview.
Arm/Group | BTDS | BTDS With Naltrexone | Naltrexone | Moxifloxacin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/66 | 0/66 | 0/66 | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 59/66 | 47/66 | 49/66 | 37/65 | 34/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BTDS (N=66) | BTDS With Naltrexone (N=66) | Naltrexone (N=66) | Moxifloxacin (N=65) | Placebo (N=65)
Infrequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 — Onset of event occurred before study drug administration.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BTDS (N=66) | BTDS With Naltrexone (N=66) | Naltrexone (N=66) | Moxifloxacin (N=65) | Placebo (N=65)
Abdominal discomfort (Gastrointestinal disorders) | 9 | 7 | 8 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 9 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 5 | 6 | 10 | 4
Flatulence (Gastrointestinal disorders) | 2 | 6 | 3 | 1 | 2
Haematochezia (Gastrointestinal disorders) | 5 | 1 | 1 | 1 | 0
Infrequent bowel movements (Gastrointestinal disorders) | 35 | 15 | 16 | 7 | 10
Nausea (Gastrointestinal disorders) | 30 | 27 | 19 | 5 | 8
Vomiting (Gastrointestinal disorders) | 16 | 9 | 7 | 1 | 4
Application site erythema (General disorders) | 6 | 5 | 8 | 8 | 2
Application site irritation (General disorders) | 10 | 5 | 5 | 5 | 9
Application site pain (General disorders) | 3 | 2 | 7 | 2 | 3
Application site papules (General disorders) | 6 | 7 | 4 | 3 | 2
Application site pruritus (General disorders) | 12 | 9 | 13 | 15 | 8
Application site rash (General disorders) | 2 | 5 | 2 | 3 | 1
Fatigue (General disorders) | 5 | 3 | 5 | 0 | 2
Feeling drunk (General disorders) | 4 | 1 | 3 | 0 | 1
Feeling hot (General disorders) | 5 | 0 | 5 | 1 | 3
Application site pustules (Infections and infestations) | 4 | 2 | 1 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 8 | 2 | 2 | 1 | 1
Dizziness (Nervous system disorders) | 18 | 8 | 7 | 2 | 4
Headache (Nervous system disorders) | 28 | 20 | 15 | 11 | 16
Somnolence (Nervous system disorders) | 7 | 5 | 2 | 0 | 1
Dysuria (Renal and urinary disorders) | 4 | 0 | 1 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days